CLINICAL TRIAL: NCT01319474
Title: Use of Whole-leg Ultrasound for Diagnosis of Deep Vein Thrombosis in Pregnant Patients
Brief Title: Whole-leg Ultrasound in Pregnant Patients
Acronym: CLOT-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Scott M. Stevens, Transitional Year Program Director, Intermountain Health Care, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 950359
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis; Pulmonary embolism; Ultrasound; Pregnancy
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound for suspected DVT (Other): Enrolled subjects suspected to have deep vein thrombosis undergo whole-leg compression ultrasound. Those with a normal result undergo clinical follow-up for thrombotic outcomes over the following three months.
  Interventions: Other: Whole-leg compression ultrasound

INTERVENTIONS:
Other: Whole-leg compression ultrasound — Duplex ultrasound assessment of the venous system of the leg(s) suspected of deep vein thrombosis. Assessment occurs from the most proximal assessable portion of the common femoral vein (usually at the inguinal ligament) to the level of the malleolus.

SUMMARY:
This study seeks to determine the rate of thromboembolic complications (blood clots), including death attributed to thromboembolic disease, when anticoagulation (blood thinner) therapy is withheld from pregnant patients suspected of deep vein thrombosis (DVT) after a whole-leg compression ultrasound shows no DVT. Patients are followed for three months after the ultrasound to determine if a blood clot is diagnosed during that time.

DETAILED DESCRIPTION:
SPECIFIC AIM To determine the rate of thromboembolic complications (including death attributed to thromboembolic disease) in pregnant patients suspected of deep vein thrombosis (DVT) when anticoagulation therapy is withheld on the basis of a negative whole-leg compression ultrasound examination (whole-leg CUS).

BACKGROUND AND SIGNIFICANCE

The diagnosis of deep vein thrombosis of the leg is challenging due to the great variability of clinical presentation and the lack of sensitivity of noninvasive tests. This is particularly true for pregnant patients, who have been excluded from most major studies of diagnostic strategies for DVT. Ironically, pregnancy is considered a major risk factor for DVT, making evidence-based diagnosis in this patient group particularly important.

A study performed at LDS Hospital, found that a single, whole-leg compression ultrasound could safely exclude the diagnosis of suspected, symptomatic, first-episode deep vein thrombosis of the leg. A subsequent metanalysis of studies of the same technique confirmed this finding, but observed that the utility of this strategy in pregnant patients required further study, as only 57 of the over 4,500 subjects in the pooled metanalysis were pregnant.

Therefore, better information regarding the performance of diagnostic testing for suspected DVT in pregnant patients is needed. If whole-leg compression ultrasound proves adequately sensitive in this patient group, this will be a significant step in simplifying the diagnostic process for deep vein thrombosis, and will confirm the diagnostic strategy most commonly used presently by physicians at Intermountain Medical Center.

EXPERIMENTAL DESIGN AND METHODS

Design Prospective clinical cohort study ("management study").

Patients 268 sequentially-enrolled pregnant patients evaluated for suspected symptomatic deep vein thrombosis of the leg, reporting to the Intermountain Medical Center Peripheral Vascular Laboratory. Vascular technicians will pre-screen patients for study entry with a simple questionnaire. Those meeting screening criteria will then be interviewed by the study coordinator to verify they meet inclusion criteria, have no reason for exclusion, and provide informed consent.

Demographic and medical history information:

Clinical information relevant to the study will be obtained from the Study Coordinator following informed consent during the initial study interview. Query of the Intermountain Healthcare electronic medical record will also be performed at entry. Relevant information will be included on a standardized Case Report Form.

Informed Consent documents, Case Report Forms and relevant source documents from the electronic medical record will be obtained, placed in a study binder and stored according to the policies of the Institutional Review Board.

Measurements:

A research clinician will perform a brief clinical assessment, including adequate information to calculate the LeFT clinical prediction score, which has been evaluated in a prior study. Patients will then proceed to performance of whole-leg compression ultrasound.

Objective Testing for Venous Thrombosis Whole-leg CUS will be performed on all patients. A standardized technique will be used for the CDU examination, which is identical to the protocol used clinically by the Intermountain Medical Center Peripheral Vascular Laboratory.

Compressibility of the veins will be assessed. The results will be categorized as normal if all imaged venous segments are fully compressible, as abnormal if a noncompressible segment is identified, or as inadequate for interpretation.

If the vascular technologist develops suspicion of isolated iliac DVT (based on absence of phasic respiratory flow or complete absence of flow in the common femoral vein by Doppler, but with normal compression) the referring physician and principal investigator will be contacted immediately by telephone. Further evaluation (usually by an alternate imaging modality) will be ordered at the discretion of the referring physician according to best clinical judgment.

Interpretation will be performed by experienced vascular surgery staff according to protocols currently in use at Intermountain Medical Center. Findings will be redacted to specific data fields by the interpreting surgeon according to a form generated for this purpose, and entered onto a Case Report Form.

Interobserver variability will be limited by using a priori criteria for a positive and negative study. Interobserver agreement for this technique has been found to be high in a prior study.

If the result of initial whole-leg CUS is normal (no DVT identified), anticoagulation will be withheld, regardless of symptoms.

If the result of testing is abnormal (DVT identified), the patient will be referred to the treating clinician for usual management at the discretion of the clinician. This group will not be followed for study outcomes.

Subjects whose results are classified as inadequate for interpretation will have reasons logged and be excluded from analysis. They will receive further management according to the discretion of the treating physician.

Long-Term Follow-up Patients with a negative whole-leg CUS will undergo three months of clinical follow-up, a strategy used in many diagnostic trials for DVT.2 Patients will be instructed to return immediately to our emergency department if they have symptoms or signs of DVT or pulmonary embolism (PE). A study clinician will assess them at 3 months by telephone interview using a standardized questionnaire.

If patients contact the study team with symptoms suspicious for DVT or PE, they will be evaluated by a study clinician in the Thrombosis Clinic (symptoms of DVT), or referred to emergent care for evaluation (symptoms of PE). Participants' treating clinicians are also free to obtain any medically appropriate diagnostic testing for suspected DVT or PE during the follow-up period. A letter will be sent to referring physicians explaining the protocol and emphasizing that any appropriate diagnostic testing for suspected DVT or PE may be performed as clinically indicated.

At the follow-up assessment, an interval history will be taken with emphasis on specific symptoms (including leg pain, tenderness and swelling, chest pain, dyspnea, hemoptysis, and syncope), hospitalization, interval evaluation for DVT or PE and use of anticoagulants. For all patients who die, the cause of death will be determined from autopsy or by independent clinical review if autopsy cannot be obtained. If at follow-up a patient identifies symptoms suspicious for DVT or PE that have not previously been clinically evaluated, they will be scheduled for an in-person evaluation with a physician in the Intermountain Medical Center Thrombosis Clinic.

In addition to information obtained from the patient during the follow-up visit, a comprehensive review of the patient's Intermountain electronic health record will be performed to look for evidence of diagnostic testing for deep vein thrombosis or pulmonary embolism or use of anticoagulant medications. Additionally, the study coordinator presently receives alerts of all positive diagnostic tests for DVT and PE performed in the facility daily. This list will be reviewed for study participants.

Results of the follow-up assessment will be entered on a Case Report Form by study staff. This form will be added to the study binder by the study coordinator and information appended to the database by the data entry clerk.

The study will be designed to estimate the event rate of thromboembolic disease and death attributable to thromboembolic disease in the normal cohort during the three-month follow-up period. An exact 95% confidence interval that excludes a rate of VTE of 3% or greater will be defined as clinically acceptable, in accordance with previous trials of DVT diagnosis.

The study will report analysis of outcomes both on a per-protocol and intention-to-treat basis in the event of protocol violation (i.e. receipt of therapeutic anticoagulation despite negative whole-leg ultrasound, without objective evidence of a thrombotic complication).

In the event of withdrawal of participation, affected subjects will be suppressed from analysis (i.e. analysis will be performed on a per protocol basis), or in the event that isolated iliac DVT is diagnosed following vascular technologist suspicion. Isolated iliac DVT diagnosed after additional imaging resulting from technologist suspicion will be analyzed as an additional outcome variable, and the rate of this diagnosis reported with a corresponding exact 95% confidence interval. Use of intention-to-treat analysis could bias results of the study in the case of withdrawn subjects as they would, by definition, not complete the defined follow-up period and would not have ascertainment of the primary study outcome.

Adjudication of Outcomes A panel of three independent physicians with established expertise in venous thromboembolism will be named to adjudicate all suspected events of DVT or PE, and all diagnostic tests for these occurring during the follow-up period. Simple majority will resolve disputes. All deaths will be adjudicated as to whether attributable to PE or another cause by the same group of adjudicators.

Methodological Issues and Avoidance of Bias Entering consecutive patients into the study will avoid selection bias. To avoid bias during the initial testing period, we have established pre-defined criteria for negative and positive studies. Further diagnostic testing on patients with negative results will not be undertaken unless dictated by new or progressive symptoms. Patients with a negative whole-leg CUS will not be treated and therapy will be given to all patients with positive results.

Diagnostic suspicion bias will be avoided by objectively testing all patients who return during follow-up with symptoms or signs suggestive of deep venous thrombosis or pulmonary embolism. Interpretation bias will be avoided by obtaining independent interpretation of follow-up testing in patients with suspected disease by independent adjudicators. The adjudicators will be blinded to the results of the initial ultrasound and the cohort to which the patient belongs. All deaths will be independently reviewed. The adjudicators will be blinded to the cohort to which the patient belongs.

Patient confidentiality will be maintained by keeping the patient identity log separate from the database, which will use only unique numerical identifiers. Complete data tracking will be assured by comparison of enrollment log and database by independent reviewer.

STATISTICAL ANALYSIS

Descriptive statistics for age, weight, height, trimester (weeks gestation), symptoms at presentation (pain, tenderness, duration of symptoms), clinical conditions (recent surgery, recent hospitalization, cancer, congestive heart failure, recent immobilization, cellulitis, superficial phlebitis and family history of thromboembolic disease) and the LeFT variables (including leg circumference) will be calculated to characterize the study population.

The event rate of thromboembolic complications and death from thromboembolic disease will be calculated for patients with negative whole-leg CUS; both per-protocol and by intention-to-treat.

The rate of isolated iliac DVT detected after vascular technologist suspicion will be reported as a separate calculation with corresponding exct 95% confidence interval

A two-sided confidence interval for the event rate (objectively verified venous thromboembolism) will be calculated for the observation cohort by exact methods. If this confidence interval excludes the commonly accepted threshold event rate of 3%, we will conclude that the diagnostic strategy is clinically valid.

We will also describe the clinical characteristics of clots (e.g. venous distribution) and other endpoints when those data are available.

The sample size of 268 patients who meet eligibility criteria was chosen so that an exact 95% confidence interval would exclude an event rate of venous thromboembolism in the observation cohort of 3%. Excluding an event rate of 3% is the commonly accepted standard by which diagnostic strategies are deemed clinically acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Be suspected by the referring medical provider to have a first episode of acute DVT of the lower extremities.
* Be presenting for the initial diagnostic ultrasound for the present symptom complex.
* Pregnancy confirmed by an objective test.
* Be > 18 years old.
* Provide written informed consent.

Exclusion Criteria:

* Compression ultrasonography cannot be performed due to physical or technical reasons.
* The patient has a prior history of DVT in the ipsilateral leg.
* Previous venous ultrasound has been performed during the same pregnancy.
* The patient is suspected by the referring clinician to have symptomatic pulmonary embolism.
* Long-term follow-up will not be possible due to geographic inaccessibility, homelessness or lack of a telephone.
* Therapeutic doses of an anticoagulant have been received for more than 24 hours before enrollment.
* Long term anticoagulation will be required for another diagnosis (e.g. atrial fibrillation).
* Informed consent cannot be obtained.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2011-02; Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptomatic VTE | Three months
  The primary outcome measure will be DVT or PE, or death attributable to thromboembolic disease confirmed by objective testing in the 3 months following enrollment.

SECONDARY OUTCOMES:
Isolated iliac DVT | At enrollment
  The exact rate of isolated iliac vein DVT identified on futher testing performed on the basis of suspicious doppler ultrasound findings.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Stevens, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermoutain Medical Center, Murray, Utah, United States

REFERENCES:
- [Background] Wells PS, Anderson DR. Modern approach to diagnosis in patients with suspected deep vein thrombosis. Haemostasis. 1999 Dec;29 Suppl S1:10-20. doi: 10.1159/000054107. PMID 10629399
- [Background] Chan WS, Lee A, Spencer FA, Crowther M, Rodger M, Ramsay T, Ginsberg JS. Predicting deep venous thrombosis in pregnancy: out in "LEFt" field? Ann Intern Med. 2009 Jul 21;151(2):85-92. doi: 10.7326/0003-4819-151-2-200907210-00004. PMID 19620161
- [Background] Stevens SM, Elliott CG, Chan KJ, Egger MJ, Ahmed KM. Withholding anticoagulation after a negative result on duplex ultrasonography for suspected symptomatic deep venous thrombosis. Ann Intern Med. 2004 Jun 15;140(12):985-91. doi: 10.7326/0003-4819-140-12-200406150-00007. PMID 15197015
- [Background] Johnson SA, Stevens SM, Woller SC, Lake E, Donadini M, Cheng J, Labarere J, Douketis JD. Risk of deep vein thrombosis following a single negative whole-leg compression ultrasound: a systematic review and meta-analysis. JAMA. 2010 Feb 3;303(5):438-45. doi: 10.1001/jama.2010.43. PMID 20124539